CLINICAL TRIAL: NCT05759065
Title: A Hybrid Effectiveness Implementation Trial Evaluating Behavioral Treatments for Insomnia for Socioeconomically Disadvantaged Adults in Primary Care
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Suzanne M. Bertisch, MD, MPH, Associate Physician, Clinical Director of Behavioral Sleep Medicine, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023P000106
Record Dates: First submitted 2023-02-08; First posted 2023-03-08 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tele-Brief Behavioral Treatment for Insomnia (Experimental)
  Interventions: Behavioral: Tele-Brief Behavioral Treatment for Insomnia
- Tele-Cognitive-Behavioral Therapy for Insomnia (Active Comparator)
  Interventions: Behavioral: Tele-Cognitive-Behavioral Therapy for Insomnia

INTERVENTIONS:
Behavioral: Tele-Brief Behavioral Treatment for Insomnia — Brief Behavioral Treatment for Insomnia (BBTI) comprises of up to five weekly intervention visits by phone, delivered by a variety of practitioners without formal training in sleep.
  Arms: Tele-Brief Behavioral Treatment for Insomnia
Behavioral: Tele-Cognitive-Behavioral Therapy for Insomnia — Cognitive-Behavioral Therapy for Insomnia (CBTI) is a multicomponent strategy delivered by trained mental health clinicians over 6 to 12 weeks.
  Arms: Tele-Cognitive-Behavioral Therapy for Insomnia

SUMMARY:
The overall objective of this study is to conduct a randomized effectiveness-implementation trial to test the non-inferiority of tele-Brief Behavioral Treatment for Insomnia vs. tele-Cognitive-Behavioral Therapy for Insomnia among socioeconomically disadvantaged adults with insomnia in the primary care setting.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Meet clinical diagnostic criteria for insomnia
* Insomnia severity score > 10
* Eligible to receive care through publicly supported medical assistance, OR
* Identify as race or ethnic minority
* Has capacity for informed consent

Exclusion Criteria:

* Untreated, current major depressive disorder
* History of bipolar or psychosis
* Active substance abuse or drug abuse
* Excessive daytime sleepiness
* Seizure within the past 1 year
* Main sleep period outside of 8pm - 11am
* Regular nightshift work
* Untreated, previously diagnosed moderate to severe sleep apnea
* Severe medical condition, which may require hospitalizations over the next 6 months
* Active suicidal ideation, if elicited passively during screening
* Pregnant or planning to become pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2024-04-02 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Insomnia severity index, ISI | 3 months
  The Insomnia Severity Index is a 7-item self-report questionnaire assessing the nature, severity, and impact of insomnia in the last month. A 5-point Likert scale is used to rate each item (e.g., 0 = no problem; 4 = very severe problem), yielding a total score ranging from 0 to 28. The total score is interpreted as follows: absence of insomnia (0-7); sub-threshold insomnia (8-14); moderate insomnia (15-21); and severe insomnia (22-28).

SECONDARY OUTCOMES:
Insomnia severity index, ISI | 6- and 12-months
  The Insomnia Severity Index is a 7-item self-report questionnaire assessing the nature, severity, and impact of insomnia in the last month. A 5-point Likert scale is used to rate each item (e.g., 0 = no problem; 4 = very severe problem), yielding a total score ranging from 0 to 28. The total score is interpreted as follows: absence of insomnia (0-7); sub-threshold insomnia (8-14); moderate insomnia (15-21); and severe insomnia (22-28).
Quality of Life and Symptoms - Patient-Reported Outcomes Measurement Information System (PROMIS) Global Health | 3-months
  The PROMIS Global Health measures assess an individual's physical, mental and social health. The measure produces two scores: Physical and Mental Health from 4 items each. Item responses are combined to yield a T-score with a population mean of 50 and standard deviation of 10.
Quality of Life and Symptoms - Generic-quality of life | 3-months
  Generic-quality of life will be assessed by the change in the Euroqol - 5 Dimensions (EQ-5D) questionnaire. The questionnaire comprises of 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, and extreme problems. There is no total score or range.
Generalized Anxiety Disorder (GAD-7) | 3-months
  GAD-7 measures self-reported anxiety disorder. The measure includes 7-items with higher scores indicating anxiety. The minimum score is 0 and the maximum score is 21.
Patient Health Questionnaire for depression (PHQ-8) | 3-months
  PHQ-8 measures self-reported current depression. The measure includes 8-items with higher scores indicating depression. The minimum score is 0 and the maximum score is 24.
Patient-Reported Outcomes Measurement Information System (PROMIS) Sleep Impairment, 8a | 3-months
  PROMIS Sleep Impairment measures self-reported perceptions of alertness, sleepiness, and tiredness during usual waking hours, and the perceived functional impairments during wakefulness associated with sleep problems or impaired alertness during the past seven days. The measure includes 8-items with higher scores indicating greater sleep impairment. The minimum score is 8 and the maximum score 40. Item responses are combined to yield a T-score with a population mean of 50 and standard deviation of 10.
Patient-Reported Outcomes Measurement Information System (PROMIS) Sleep Disturbance, 8b | 3-months
  PROMIS Sleep Disturbance measures self-reported sleep quality and associated daytime functioning during the past seven days. The measure includes 8-items with higher scores indicating greater sleep disturbance. The minimum score is 8 and the maximum score is 40. Item responses are combined to yield a T-score with a population mean of 50 and standard deviation of 10.
Diary reported sleep duration | 3-months
  Self-reported sleep duration with be measured using sleep diary
Diary-reported sleep efficiency | 3-months
  Self-reported sleep efficiency with be measured using sleep diary
Number of participants with hypnotic use self-reported from the sleep diary | 3-months
  Hypnotic use will be measured by the number of participants who self-reported use on the sleep diary

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No